CLINICAL TRIAL: NCT03458689
Title: Quadratus Lumborum Block Versus Transversus Abdominis Plane Block in Patients Undergoing Left Hemicolectomy: A Randomized Controlled Trial
Brief Title: Quadratus Lumborum Block Versus Transversus Abdominis Plane Block in Patients Undergoing Left Hemicolectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ostfold Hospital Trust (Other)
Responsible Party: Principal Investigator, Jan Sverre Vamnes, Senior conultant, Ph.D., Ostfold Hospital Trust
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 1813
Record Dates: First submitted 2018-02-28; First posted 2018-03-08 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Colon Neoplasm; Surgery; Pain, Postoperative
MeSH Terms: conditions — Colonic Neoplasms; Pain, Postoperative | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant
Masking Description: Information connecting the patients to the data are kept locked and will be destroyed after the end of the investigation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Left hemicolectomy without nerve blocks (Other): Left hemicolectomy, laparoscopic technique Enteral and parenteral analgesics such as paracetamol and oksykodon
  Interventions: Procedure: Left hemicolectomy, laparoscopic technique
- Left hemicolectomy with TAP block (Active Comparator): Left hemicolectomy, laparoscopic technique TAP block bilateral with Naropin 3,75 mg/ml, 2 x 20 ml
  Interventions: Procedure: Left hemicolectomy, laparoscopic technique
- Left hemicolectomy with QL block (Active Comparator): Left hemicolectomy, laparoscopic technique QL block bilateral with Naropin 3,75 mg/ml, 2 x 20 ml
  Interventions: Procedure: Left hemicolectomy, laparoscopic technique

INTERVENTIONS:
Procedure: Left hemicolectomy, laparoscopic technique — Left hemicolectomy, Laparoscopic technique
  Other Names: QL block bilateral with ropivacain 3,75 mg/ml (2 x 20 ml); TAP block with ropivacain 3,75 mg/ml (2 x 20 ml); Traditional analgesics such as paracetamol and oksycodon

SUMMARY:
The enhanced recovery after surgery and laparoscopic approach have been proven beneficial in surgery of the colon. However, patients have still pain, nausea and vomiting postoperatively. Postoperative pain is an expected but undesirable effect after an operation. This study will compare Transabdominis Plane (TAP) Block and Quadratus Lumborum (QL) Block with the common postoperative treatment with enteral and parenteral analgesics.

DETAILED DESCRIPTION:
TAP is a recommended multimodal method of reducing postoperative pain in laparoscopic and open surgery. TAP block seems to be feasible and effective in postoperative pain control without increasing morbidity in colon resections. QL block is also performed as one of the perioperative pain management procedures in abdominal surgery. It is regarded as an effective analgesic tool. The dermatomal effects of QL block reach higher than the TAP block, and might explain the better effect of the QL block than TAP blocks on postoperative pain after caesarean delivery. For this study the investigators standardize the type of surgery to be left hemicolectomy. This is the most common procedure on colon.

Power and Sample Size Calculator:

The number of patients required for the study was calculated on the basis of opioid consumption. We were interested in a reduction by 20% in the group given QLB. Assuming α=0,05, we calculated that we need 69 patients (23 in each group) to achieve a power of 80% (β=0.2).

75 adult patients scheduled for left hemicolectomy have to be included.

Subcutaneous wound infiltration at the end of surgery in all patients with ropivacaine 2 mg/ml, 20 ml. Maximum allowed dosis of Ropivacain is 3 mg/kg bodyweight (BW), dosis reduction if BW<70 kg Premedication: Paracetamol 2 g and Diklofenak 100 mg orally. General anaesthesia: TCI: Propofol and Remifentanil Ondansetron 4 mg, dexamethasone 8 mg and Oxycodone 5 mg intravenously at the end of surgery.

Postoperatively:

Oral paracetamol and codeine-fixed combination up to 1000 mg and 60 mg, respectively, every 6 h In case of insufficient analgesia, as judged by the patient, oxycodon 2 - 5 mg IV.

When nausea and vomiting occure postoperatively, ondansetron 4 mg IV administers as the drug of first choice followed by droperidol 0,625 mg IV if the nausea/vomiting persists.

Collected data:

Postoperative pain at rest and during activity evaluated by a 4-points verbal pain score (VPS; with no pain=0, slight pain = 1, Moderate pain = 2, and severe pain = 3) on admission to recovery, and every hour until discharge.

Rescue analgesic consumption during 0 to 4, 4 to 24 and 24 to 48 h. Sedation, nausea and vomiting record by the same 0 - 3 scale (none, slight, moderate, strong) during recovery Time of postoperative mobilization with corresponding pain score. Time of discharge-to-home or ward readiness according to standard criteria, including stable vital signs, no bleeding from the surgical site, ability to void, absence of excessive nausea and pain, and ability to dress and walk without support.

Side effects including nausea and/or vomiting (0 to 4, 4 to 24, and 24 to 48 h), antiemetics administered (0 to 24 and 24 to 48 H), grade of sedation (0 to 10 scale, where 0 = awake, and 10 = aroused on stimulation), and other side effects and symptoms of LA toxicity.

Telephone interview at 24 h, 48 h and 7 days, with questions:

Pain during rest and activity using the VPS Total need of analgesics Sedation Nausea Level of activity Overall satisfaction with the per- and postoperative period on a 0 - 3 scale: not satisfied, slight, moderate or highly satisfied.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 Years
* BMI 20-35
* ASA physical status I-II

Exclusion Criteria:

* Allergy to LA
* Chronic pain requiring opioid analgesics
* Patients with atrioventricular block II
* Patients treated with class III antiarrhythmics
* Patients with severe renal and/or hepatic disease
* A coagulation disorder
* An infection at the LA injection place

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2018-02-28 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Use of analgesics - "change" is being assessed | 1 week (0-4 hrs) (4-24 hrs) (24-48 hrs) (48 - 168 hrs)
  Amount of analgesics used postoperative

SECONDARY OUTCOMES:
Pain at the incision site - "change" is being assessed | 1 week (0-4 hrs) (4-24 hrs) (24-48 hrs) (48 - 168 hrs)
  VPS (Verbal Pain Score): No pain = 0, Slight pain = 1, Moderate pain= 2, Severe pain = 3
Deep pain and pain on coughing - "change" is being assessed | 1 week (0-4 hrs) (4-24 hrs) (24-48 hrs) (48 - 168 hrs)
  VPS (Verbal Pain Score): No pain = 0, Slight pain = 1, Moderate pain= 2, Severe pain = 3
Nonsteroidal anti-inflammatory drug consumption - "change" is being assessed | 1 week (0-4 hrs) (4-24 hrs) (24-48 hrs) (48 - 168 hrs)
  Amount of different medicaments in mg
Postoperative nausea and vomiting - "change" is being assessed | 1 week (0-4 hrs) (4-24 hrs) (24-48 hrs) (48 - 168 hrs)
  0 - 3 score where None = 0, Little nausea = 1, Can not eat = 2, Vomiting = 3
Antiemetic administered - "change" is being assessed | 1 week (0-4 hrs) (4-24 hrs) (24-48 hrs) (48 - 168 hrs)
  Amount of different medicaments in mg
Sedation scores - "change" is being assessed | 1 week (0-4 hrs) (4-24 hrs) (24-48 hrs) (48 - 168 hrs)
  Sleepy or active. Score: Awake = 0, Tired = 1, Falls asleep = 2, Asleep all the time = 3

CONTACTS AND LOCATIONS:
Overall Officials: Jan Sverre Vamnes, MD, Ph.D., Principal Investigator — Senior Consultant
Locations (1):
- Ostfold Hospital Trust, Moss, Grålum, Østfold fylke, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Borglum J, Gogenur I, Bendtsen TF. Abdominal wall blocks in adults. Curr Opin Anaesthesiol. 2016 Oct;29(5):638-43. doi: 10.1097/ACO.0000000000000378. PMID 27429253
- [Result] Blanco R, Ansari T, Riad W, Shetty N. Quadratus Lumborum Block Versus Transversus Abdominis Plane Block for Postoperative Pain After Cesarean Delivery: A Randomized Controlled Trial. Reg Anesth Pain Med. 2016 Nov/Dec;41(6):757-762. doi: 10.1097/AAP.0000000000000495. PMID 27755488
- [Result] El-Dawlatly AA, Turkistani A, Kettner SC, Machata AM, Delvi MB, Thallaj A, Kapral S, Marhofer P. Ultrasound-guided transversus abdominis plane block: description of a new technique and comparison with conventional systemic analgesia during laparoscopic cholecystectomy. Br J Anaesth. 2009 Jun;102(6):763-7. doi: 10.1093/bja/aep067. Epub 2009 Apr 17. PMID 19376789
- [Result] Murouchi T, Iwasaki S, Yamakage M. Quadratus Lumborum Block: Analgesic Effects and Chronological Ropivacaine Concentrations After Laparoscopic Surgery. Reg Anesth Pain Med. 2016 Mar-Apr;41(2):146-50. doi: 10.1097/AAP.0000000000000349. PMID 26735154
- [Result] Pirrera B, Alagna V, Lucchi A, Berti P, Gabbianelli C, Martorelli G, Mozzoni L, Ruggeri F, Ingardia A, Nardi G, Garulli G. Transversus abdominis plane (TAP) block versus thoracic epidural analgesia (TEA) in laparoscopic colon surgery in the ERAS program. Surg Endosc. 2018 Jan;32(1):376-382. doi: 10.1007/s00464-017-5686-7. Epub 2017 Jul 1. PMID 28667547
- [Result] Ueshima H, Otake H, Lin JA. Ultrasound-Guided Quadratus Lumborum Block: An Updated Review of Anatomy and Techniques. Biomed Res Int. 2017;2017:2752876. doi: 10.1155/2017/2752876. Epub 2017 Jan 3. PMID 28154824